CLINICAL TRIAL: NCT02353468
Title: Phase II Study: Therapy With Bortezomib + Lenalidomide + Dexamethasone With Lenalidomide + Dexamethasone as Post Transplant Consolidation and Maintenance for Patients With Symptomatic Multiple Myeloma Following Autologous Transplantation
Brief Title: Bortezomib, Lenalidomide, and Dexamethasone in Treating Patients With Multiple Myeloma Undergoing Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principle investigator left the institution
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0816.cc; NCI-2011-03113 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-01

CONDITIONS: Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzyme inhibitor, biological therapy, chemotherapy (Experimental): CONSOLIDATION: Patients receive VLD therapy comprising bortezomib IV on days 1, 4, 8, and 11, lenalidomide PO QD on days 1-14, and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Courses continue for 28 days and repeat every 3 months in the absence of disease progression or unacceptable toxicity.
  In between courses of VLD, patients receive LD therapy comprising lenalidomide PO QD on days 1-21 and dexamethasone PO QD or IV every Monday (x3). Courses continue for 28 days.
  MAINTENANCE: Starting in the third year of therapy, patients receive lenalidomide PO QD on days 1-14 and dexamethasone PO QD or IV every Monday (x2). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: Velcade
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; IMiD-1
Drug: Dexamethasone — Given PO or IV
  Other Names: Decadron

SUMMARY:
This phase II trial studies how well giving bortezomib, lenalidomide, and dexamethasone together works in treating patients with multiple myeloma undergoing stem cell transplant. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib, lenalidomide, and dexamethasone together may kill more cancer cells.

DETAILED DESCRIPTION:
CONSOLIDATION: Patients receive bortezomib, lenalidomide, and dexamethasone (VLD) therapy comprising bortezomib intravenously (IV) on days 1, 4, 8, and 11, lenalidomide orally (PO) once daily (QD) on days 1-14, and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Courses continue for 28 days and repeat every 3 months in the absence of disease progression or unacceptable toxicity.

In between courses of VLD, patients receive Lenalidomide + Dexamethasone (LD) therapy comprising lenalidomide PO QD on days 1-21 and dexamethasone PO QD or IV every Monday (x3). Courses continue for 28 days.

MAINTENANCE: Starting in the third year of therapy, patients receive lenalidomide PO QD on days 1-14 and dexamethasone PO QD or IV every Monday (x2). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic active multiple myeloma who have completed autotransplant are eligible for the study; patients should be assessed for eligibility within 35 days of the transplant and treatment should commence within 10 weeks of the transplant
* Performance status of 0-2 based on Southwest Oncology Group (SWOG) criteria; patients with a poor performance status (3-4) are also eligible, if complications of the bone such as compression fracture, hyperviscosity or infection such as pneumonia have been adequately treated
* No significant co-morbid medical conditions; no uncontrolled life threatening infection
* Unsupported platelet count > 80,000/uL
* Absolute neutrophil count (ANC) > 1000/uL
* Signed informed consent should be obtained from all patients in accordance with institutional and federal guidelines

Exclusion Criteria:

* Patients with a history of recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, difficult to control significant cardiac arrhythmias, or arrhythmia associated with prolonged QT interval
* Pregnant or nursing women; women of child-bearing potential must have a negative pregnancy documented within one week of registration; women/men of reproductive potential may not participate unless they have agreed to use two forms of effective contraceptive method
* Patients with a grade 3-4 neuropathy related to prior exposure to bortezomib, thalidomide, or other agents
* Human immunodeficiency virus (HIV) positive patients
* Transaminases > 2 x normal values
* Bilirubin > 2 x normal values
* Active uncontrolled infection
* History of significant psychiatric illness; steroid induced psychosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Choon-kee Lee, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2009 and October 2011, 3 patients were enrolled in the study from University of Colorado Cancer Center
Pre-assignment Details: 35 days following autologous transplant, patients were evaluated for eligibility by the standard tests, including paraprotein assessment, bone marrow biopsy and aspiration, MRI scan, and PET/CT scan that is indicated for patients with hypo- or non-secretary myeloma.
Groups:
- Enzyme Inhibitor, Biological Therapy, Chemotherapy: CONSOLIDATION: Patients received VLD therapy comprising bortezomib IV on days 1, 4, 8, and 11, lenalidomide PO QD on days 1-14, and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Courses continue for 28 days and repeat every 3 months in the absence of disease progression or unacceptable toxicity.
  In between courses of VLD, patients received LD therapy comprising lenalidomide PO QD on days 1-21 and dexamethasone PO QD or IV every Monday (x3). Courses continue for 28 days.
  MAINTENANCE: Starting in the third year of therapy, patients received lenalidomide PO QD on days 1-14 and dexamethasone PO QD or IV every Monday (x2). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Lenalidomide: Given PO
  Dexamethasone: Given PO or IV
Period: Overall Study
Arm/Group | Enzyme Inhibitor, Biological Therapy, Chemotherapy
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated | 3

BASELINE CHARACTERISTICS:
Population: The study had planned to enroll sixty-two patients in order to achieve sufficient power, 81% to detect an improvement in 3-year event-free survival.
Arm/Group | Enzyme Inhibitor, Biological Therapy, Chemotherapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Rates by Land-mark Analysis
Description: A Kaplan-Meier curve would have been used to describe the distribution.
Time Frame: up to 5 years
Population: The study was terminated, study endpoints were not reached.
Arm/Group | Enzyme Inhibitor, Biological Therapy, Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events for approximately 2 years until the study was terminated.
Arm/Group | Enzyme Inhibitor, Biological Therapy, Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study was terminated due to the investigator's departure from the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes